CLINICAL TRIAL: NCT06281067
Title: Reassessment of myocardIAL Bridge TOwards PeRsOnalized Medicine: RIALTO PRO
Brief Title: Reassessment of myocardIAL Bridge TOwards PeRsOnalized Medicine
Acronym: RIALTO PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Domenico D'Amario, Prof, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 271.673
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Bridge
Keywords: myocardial bridge; Personalized Medicine
MeSH Terms: conditions — Myocardial Bridging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "full-physiology approach" arm (Experimental): In the "full-physiology approach" arm, patients will be, during CA, simultaneously subjected to a full interventional diagnostic procedure, including:
  * resting distal coronary pressure to aortic pressure ratio (Pd/Pa);
  * fractional flow reserve (FFR) after intravenous adenosine administration;
  * Resting Ful-Cycle Ratio (RFR);
  * coronary flow reserve (CFR) and index of microvascular resistance (IMR);
  * assessment of FFR, CFR and IMR after inotropic stimulation with dobutamine (respectively FFR-d, CFR-d and IMR-d);
  * acetylcholine (ACH) provocative test.
  Interventions: Diagnostic Test: "full-physiology approach" arm
- "standard approach" arm (Other): In the "standard approach" arm, patients will undergo only an angiographic evaluation, without any invasive intracoronary assessment.
  Interventions: Diagnostic Test: "standard approach" arm

INTERVENTIONS:
Diagnostic Test: "full-physiology approach" arm — * All MB patients belonging to the full-physiology arm will undergo functional assessment of the intramural artery with basal Pd/Pa, FFR (after intravenous adenosine), RFR, CFR and IMR.
  * In the presence of a negative functional assessment (Pd/Pa> 0.92, FFR> 0.80, RFR> 0.89, CFR≥ 2.0 and IMR< 25), FFR, CFR and IMR will be measured after inotropic stimulation with dobutamine (respectively FFR-d, CFR-d and IMR-d) to exalt the epicardial hemodynamic significance of MB or its impact on structural microvascular remodelling (impaired endothelium-independent vasodilatation).
  * In the absence of epicardial hemodynamic significance (FFR-d> 0.75) and structural microvascular dysfunction (CFR≥ 2.0 and IMR< 25), ACH provocative test will be performed to evaluate the presence of epicardial or microvascular spasm (impaired endothelium-dependent vasodilatation).
  Arms: "full-physiology approach" arm
Diagnostic Test: "standard approach" arm — In the "standard approach" arm patients will undergo an angiographic evaluation of the tunnelled artery
  Arms: "standard approach" arm

SUMMARY:
The "RIALTO-PRO" study aims to optimize the diagnostic and therapeutic algorithm for myocardial bridge (MB) patients, testing the diagnostic value of a full invasive diagnostic procedure, and, consequently, the prognostic value of a tailored approach. the study objective is to determine the diagnostic and prognostic value of a full-physiology approach strategy versus a standard approach strategy in patients with a MB.

The "RIALTO PRO" study is a randomized, multicentre, prospective, open-label, superiority trial comparing a personalised versus standard management in patients with MB. Consenting and eligible patients will be randomised 1:1 to either a "full-physiology approach", consisting of a comprehensive diagnostic algorithm aimed at unmasking the main pathophysiological mechanism of myocardial ischemia and consequently a tailored treatment, or a "standard approach", consisting of angiographic evaluation of the tunnelled segment.

DETAILED DESCRIPTION:
TRIAL PROCEDURES Once MB is angiographically detected, eligible and consenting patients will be randomly assigned in a 1:1 ratio to receive a "standard approach" or a "full-physiology approach" during index CA.

Index coronary angiography Coronary angiography will be performed through a radial or femoral approach. Unfractionated heparin (initial weight-adjusted intravenous bolus of 50-70 IU/kg, with repeat boluses to achieve an activated clotting time ∼250) will be administered in all patients. To fully expose all segments of the coronary arteries, at least 2 perpendicular projections for the right coronary artery (RCA) and 4 projections for the LAD will be taken. Intracoronary nitrates can be used (depending on blood pressure and, in any case, at the discretion of the Investigator) to increase the angiographic sensitivity in detecting the "milking effect".

Physiological epicardial and microvascular assessment MB hemodynamic assessment will be performed using a diagnostic guidewire placed in the index vessel. Intravenous heparin (50-70 U/kg) should be administered to achieve therapeutic anticoagulation (activated clotting time ∼250 s). The innovative Abbott PressureWire™ X Guidewire will be used to measure pressure and temperature. The guidewire's wireless measurements are connected to an advanced platform (Coroventis‡ CoroFlow‡ Cardiovascular System) to measure physiological indices. Abbott's PressureWire™ X Guidewire and Coroventis‡ CoroFlow‡ Cardiovascular System are, nowadays, the only solution for the cath lab able to assess both epicardial vessel (i.e., FFR< 0.80) and microcirculation (i.e., CFR< 2.0 and IMR≥ 25).

Epicardial assessment will include:

* Resting Pd/Pa (n.v. > 0.92)
* FFR after intravenous adenosine administration (n.v. > 0.80)
* RFR (n.v. > 0.89)
* FFR after intravenous dobutamine administration (n.v. > 0.75) FFR is defined as the mean distal pressure (Pd)/mean aortic pressure (Pa) across MB during maximal hyperemia, achieved by administration of intravenous (140 μg/kg/min) or intracoronary bolus (up to 200 µg) of adenosine. Pd/Pa was automatically calculated by current computational software as the ratio found in the pressure recording. A cut-off of 0.80 will be used to detect hemodynamic relevance. Inotropic stimulation to exalt the hemodynamic significance of MB will be performed with intravenous dobutamine infusion, in case of a negative functional assessment (Pd/Pa> 0.92, FFR> 0.80, RFR> 0.89). The infusion will be started at 5 μg/kg/min and increased by 5μg/kg/min every 5 minutes up to 20 μg/kg/min or until the patient develops symptoms or clear evidence of ischemia. An intravenous infusion of 1 mg atropine will be administered if the patient will not experience symptoms or signs of myocardial ischemia with 20 μg/kg/min of dobutamine infusion. An intravenous bolus of β-blocker (i.e., metoprolol 5 mg) will be administered at the end of the procedure to antagonize the effects of dobutamine.

Microvascular assessment will include:

* basal CFR (n.v. ≥ 2.0) and CFR after intravenous dobutamine administration (CFR-d)
* basal IMR (n.v. < 25) and IMR after intravenous dobutamine administration (IMR-d) The coronary flow reserve and the microcirculatory resistance will be calculated using thermodilution thanks to the PressureWire™ X Guidewire. The thermodilution-based CFR cut-off value is 2.0. It is the ratio of the maximal or hyperemic flow down a coronary vessel to the resting flow. IMR is calculated as the product of distal coronary pressure at maximal hyperaemia multiplied by the hyperaemic mean transit time. Reduced CFR (< 2.0) and increased IMR (≥ 25) are representative of structural microvascular dysfunction (impaired endothelium-independent vasodilatation).

ACH provocative test In order to unmask MB-related epicardial and/or microvascular CAS, ACH provocative test will be performed in case of absence of epicardial hemodynamic significance and structural microvascular dysfunction. Incremental doses of 20, 50, 100 and 200 μg of ACH will be infused over a period of 2 minutes into the index vessel (vessel with angiographic "milking effect") via the angiographic catheter, repeating CA after each Ach dose. The test will be performed with a continuous monitoring of symptoms, electrocardiogram (ECG), and angiographic evidence of spasm. Angiographic responses during the provocation test will be assessed in multiple orthogonal views to detect the artery spasm. If either complications and/or a positive response occurred, the test will be discontinued, and higher doses will be not administered. The test will be considered positive for epicardial CAS in the presence of focal or diffuse epicardial coronary diameter reduction ≥90% in comparison with the relaxed state following intracoronary nitroglycerine administration given to relieve the spasm, associated with the reproduction of the patient's anginal symptoms and ischemic ECG shifts. Microvascular spasm will be diagnosed when typical ischemic ST-segment changes and angina develop in the absence of epicardial coronary constriction (< 90% diameter reduction). Patients who will not experience angina, spasm, or ST-segment shifts will be considered to have a negative test response (normal coronary vasoreactivity). Similarly, patients who will experience ischemic ECG shifts without angina or patients with chest pain without ischemic ECG shifts will be considered to have a negative test response.

Statistical analysis Statistical analysis will be performed using statistical software package Statistic for Data Analysis Stata 17 (64 bit; StataCorp, College Station, TX) and GraphPad Prism version 8.0.2 (GraphPad Software, San Diego, CA). Chi-square, Fisher's exact test and Kruskal Wallis test will be used to compare categorical variables. Continuous variables were listed as mean ± standard deviation (SD) and will be compared between groups using the Student's t-test, the Mann-Whitney U test, as appropriate. We will perform a 2-tailed analysis and consider a p-value ≤0.05 to be significant. With respect to the primary endpoint, all events occurring from randomization to the study end date will be counted. The number and rate of patients experiencing a primary endpoint will also be summarized. The proportion of patients remaining event-free over time will be displayed in the form of survival curves using the Kaplan-Meier method and analyzed using the log-rank test and the Gehan-Breslow-Wilcoxon test. With respect to secondary endpoints, a Cox proportional hazards model will be used, and estimates of the hazard ratios and their confidence intervals will be provided. In general, missing values will remain as missing, i.e., no attempt will be made to impute missing values and only observed values will be used in data analyses. An interim analysis will be performed on the primary endpoint when 50% of patients will have been randomized and completed the 6 months follow-up. The interim analysis will be performed by an independent statistician, blinded for the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent to the study.
2. Age ≥ 18 years and ≤ 75 years.
3. Diagnosis of MB during index coronary angiography*.
4. Symptoms or signs of inducible ischemia (if signs, these should involve the territory of the index vessel).

Angiographic definition of MB *

Myocardial bridge is a congenital anomaly characterized by an intramural course of an epicardial coronary segment. This anatomical arrangement causes the artery to be squeezed during systole, with a relaxation in diastole. In this study, MB is defined as a visual ≥ 50% reduction in the minimal luminal diameter during systole and a complete or partial relaxation in diastole ("milking effect").

The use of intracoronary vasodilators (i.e., nitrates) can increase the systolic narrowing of the vessel, through a reflex rise of the adrenergic drive, and consequently the angiographic sensitivity in detecting MB.

Exclusion Criteria:

1. Moderate to severe CAD (≥ 50% stenosis in any vessel, including chronic total occlusion) at the time of enrolment/randomization.
2. Previous CABG involving the index vessel.
3. Severe valvular heart disease.
4. Left ventricular systolic dysfunction [ejection fraction (EF) < 40%], regardless of the etiology.
5. Clinically significant right ventricular dysfunction.
6. Known severe renal impairment (eGFR < 30 ml/min/1.73 m2).
7. Known severe hepatic impairment, or history of cirrhosis with evidence of portal hypertension.
8. History of malignancy of any organ system with a life expectancy < 1 year.
9. Any previous history of ischemic stroke, intracranial haemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
10. Pregnant or breastfeeding women.
11. Known hypersensitivity or contraindication to any of the drugs used for coronary physiology testing (nitrates, adenosine, dobutamine, acetylcholine).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The composite of significant angina and MACE | at 1-year follow-up
  Composite of significant anginal burden, defined as Seattle angina questionnaire (SAQ) Summary Score ≤ 70, and MACE, defined as the composite of cardiac death, myocardial infarction, cardiac hospitalization (any cause) and target vessel revascularization at 1 year follow-up.

SECONDARY OUTCOMES:
Rate of patients with significant angina (SAQ Angina Summary Score ≤ 70) | at 1-year follow-up
Incidence of MACE | at 1-year follow-up
Rate of cardiac death | at 1-year follow-up
Rate of MI | at 1-year follow-up
Rate of cardiac hospitalization | at 1-year follow-up
Rate of TLR | at 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Patti, Prof, Study Chair — Università degli Studi del Piemonte Orientale Amedeo Avogadro
Locations (34):
- Italy (34):
  - Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale San Donato, Arezzo
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale degli Infermi di Biella, Biella
  - Policlinico S. Orsola IRCCS Azienda Ospedaliero Universitaria, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale Sant'Anna e San Sebastiano, Caserta
  - Villa Maria Cecilia Hospital, Cotignola
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria Policlinico San Martino, Genova
  - Ospedale Della Misericordia, Grosseto
  - Centro Cardiologico Monzino IRCCS, Milan
  - IRCCS Ospedale Galeazzi, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - AOU Maggiore della Carità, Novara
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale San Jacopo, Pistoia
  - Ospedali Riuniti di Rivoli, Rivoli
  - Aurelia Hospital, Roma
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Azienda Ospedaliero Universitaria Sant'Andrea, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Ospedale Sandro Pertini, Roma
  - Ospedale Santo Spirito, Roma
  - Policlinico Universitario Tor Vergata Fondazione PTV, Roma
  - Ospedale Civile Santissima Annunziata, Sassari
  - Azienda Sanitaria Provinciale di Siracusa, Syracuse
  - Azienda Ospedaliera Ordine Mauriziano, Torino
  - Azienda Ospedaliero Universitaria Città Della Salute E Scienza, Torino
  - Presidio Ospedaliero Sant'Andrea, Vercelli
  - Azienda Ospedaliera Universitaria Integrata, Ospedale Borgo Trento, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Amario D, Ciliberti G, Restivo A, Laborante R, Migliaro S, Canonico F, Sangiorgi GM, Tebaldi M, Porto I, Andreini D, Vergallo R, Leone AM, Gervasi S, Cammarano M, Palmieri V, Burzotta F, Trani C, Zeppilli P, Crea F; RIALTO Registry Investigators. Myocardial bridge evaluation towards personalized medicine: study design and preliminary results of the RIALTO registry. Eur Heart J Suppl. 2022 Nov 11;24(Suppl H):H48-H56. doi: 10.1093/eurheartjsupp/suac059. eCollection 2022 Nov. PMID 36382004
- [Background] Ciliberti G, Laborante R, Di Francesco M, Restivo A, Rizzo G, Galli M, Canonico F, Zito A, Princi G, Vergallo R, Leone AM, Burzotta F, Trani C, Palmieri V, Zeppilli P, Crea F, D'Amario D. Comprehensive functional and anatomic assessment of myocardial bridging: Unlocking the Gordian Knot. Front Cardiovasc Med. 2022 Nov 8;9:970422. doi: 10.3389/fcvm.2022.970422. eCollection 2022. PMID 36426224
- [Background] Cappannoli L, Ciliberti G, Restivo A, Palumbo P, D'Alo F, Sanna T, Crea F, D'Amario D. 'Here comes the story of the Hurricane': a case report of AL cardiac amyloidosis and myocardial bridging. Eur Heart J Case Rep. 2022 May 31;6(7):ytac225. doi: 10.1093/ehjcr/ytac225. eCollection 2022 Jul. PMID 35854894
- [Background] Montone RA, Gurgoglione FL, Del Buono MG, Rinaldi R, Meucci MC, Iannaccone G, La Vecchia G, Camilli M, D'Amario D, Leone AM, Vergallo R, Aurigemma C, Buffon A, Romagnoli E, Burzotta F, Trani C, Crea F, Niccoli G. Interplay Between Myocardial Bridging and Coronary Spasm in Patients With Myocardial Ischemia and Non-Obstructive Coronary Arteries: Pathogenic and Prognostic Implications. J Am Heart Assoc. 2021 Jul 20;10(14):e020535. doi: 10.1161/JAHA.120.020535. Epub 2021 Jul 14. PMID 34259010
- [Background] D'Amario D, Cammarano M, Quarta R, Casamassima F, Restivo A, Bianco M, Palmieri V, Zeppilli P. 'A bridge over troubled water': a case report. Eur Heart J Case Rep. 2021 Mar 31;5(3):ytab109. doi: 10.1093/ehjcr/ytab109. eCollection 2021 Mar. PMID 33824938